CLINICAL TRIAL: NCT03966352
Title: Family Building Decisions for Gay Men
Brief Title: Pathways to Fatherhood
Status: Completed | Type: Observational
Sponsor: Reproductive Medicine Associates of New Jersey (Other)
Responsible Party: Sponsor
Other Study IDs: RMA-2019-04
Record Dates: First submitted 2019-05-24; First posted 2019-05-29 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: Family Research
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — Enrolled subjects will complete a questionnaire to ascertain information on treatment considerations, obstacles, motivations, and outcomes encountered on their pathway to fatherhood.

SUMMARY:
The purpose of this study is to better understand the decision-making process that gay couples go through in order to have children.

DETAILED DESCRIPTION:
The purpose of this study is to better understand treatment considerations, obstacles, motivations, and outcomes for gay men through a survey based questionnaire study.

ELIGIBILITY:
Inclusion Criteria:

* Men over age 18 who self-identify as gay
* Participants should be individuals who are seeking or have sought reproductive services at RMA New Jersey locations.
* Participants may be included if they have not yet gone through the assisted reproductive process but are considering fatherhood and identify as gay.

Exclusion Criteria:

* Individuals who are not 18 years of age or older.
* Participants who do not self-identify as gay males.
* Female patients.
* Failure of the participant to agree to enrollment in the study with written consent.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Men who self-identify as gay
Study Population: Gay men who sought or are currently seeking family building services at an infertility practice through third party reproduction
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2019-05-24 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Response to survey questions | 1 week
  assess response to questions regarding quality of life, general health, demographic info as well as vies on sperm, egg donation, gestational carriers, legal and financial issues as well as adoption or foster care

CONTACTS AND LOCATIONS:
Locations (1):
- Reproductive Medicine Associates of New Jersey, Basking Ridge, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No